CLINICAL TRIAL: NCT03413111
Title: Modified Double Wire Technique to Facilitate the Successful Cannulation: Prospective Randomized Study
Brief Title: Modified Double Wire Technique to Facilitate the Successful Cannulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associate Professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KY20180081-1
Record Dates: First submitted 2018-01-17; First posted 2018-01-29 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-02

CONDITIONS: Biliary Cannulation; Endoscopic Retrograde Cholangiopancreatography
Keywords: ERCP; double guidewire technique

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified double wire technique (Experimental): A sphincterotome was used for standard wire-guided cannulation. If the difficult biliary cannulation occurred and guidewire inadvertently entered PD, a tiny cut of opening, with the length of 5mm, was performed with the sphincterotome. Then the guidewire was left in PD and the sphincterotome withdrew. The same sphincterotome was re-inserted in the working channel alongside the first guidewire, another wire is used for wire-guided selective cannulation of CBD. If the cannulation of CBD was not successful within 5 attempts, other cannulation techniques (e.g. transpancreatic precut, needle knife (NK) precut or over-the stent precut) would be tried at the discretion of endoscopists. A 5Fr, unflanged PD stent was placed before the ending of ERCP.
  Interventions: Procedure: Modified double wire technique
- Standard double wire technique (No Intervention): A sphincterotome was used for standard wire-guided cannulation. If the difficult biliary cannulation occurred and guidewire inadvertently entered PD, the guidewire was left in PD and the sphincterotome withdrew. The same sphincterotome was re-inserted in the working channel alongside the first guidewire, another wire is used for wire-guided selective cannulation of CBD. If the cannulation of CBD was not successful within 5 attempts, other cannulation techniques (e.g. transpancreatic precut, NK precut or over-the stent precut) would be tried at the discretion of endoscopists. A 5Fr, unflanged PD stent was placed before the ending of ERCP.

INTERVENTIONS:
Procedure: Modified double wire technique — For experimental arm, a tiny cut of papilla orifice, with the length of 5mm, was performed by sphincterotome before the double wire cannulation.
  Arms: Modified double wire technique

SUMMARY:
Selective cannulation is considered the most challenging step for most of Endoscopic retrograde cholangiopancreatography (ERCP). Wire-guided cannulation is the standard technique for initial cannulation. When meeting difficulty, double wire technique (DWT) is widely used. With one guidewire occupying pancreatic duct (PD), the following cannulation of common bile duct (CBD) with a sphincterotome preloaded with another guidewire often becomes feasible. However, because of the small opening of the papilla, sometimes it is technically challenging for the following cannulation of CBD with the sphincterotome and PD guidewire in the same working channel. We hypothesized that a tiny cut of the opening of papilla, without the injury of pancreatic sphincter, may facilitate the success of DWT and shorten the overall cannulation time.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-90 with native papilla;
* CBD as the targeted duct;
* Inadvertent PD cannulation more than twice;
* Selective biliary cannulation was not possible within 10 minutes or 5 attempts.

Exclusion Criteria:

* Contraindications of ERCP;
* Major or minor PD as the targeted duct;
* NK or transpancreatic precut before enrollment ;
* Surgically altered GI anatomy;
* Papillary carcinoma or stone impaction within papilla or fistula in papilla;
* Prior endoscopic sphincterotomy;
* Complete pancreas divisum;
* failure of pancreatic duct cannulation;
* Pregnant or breastfeeding women;
* Unwilling or inability to provide consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-02-02 (Actual); Primary Completion 2019-01-16 (Estimated); Study Completion 2019-02-16 (Estimated)

PRIMARY OUTCOMES:
Success rate of double wire technique | 3 hours
  the rate of successful cannulation of CBD for ≤5 attempts by using the sphincterotome alongside the PD guidewire.

SECONDARY OUTCOMES:
cannulation time of double wire technique | 3 hours
  the time taken from the touching of papilla by the sphincterotome alongside the PD guidewire to the successful cannulation of CBD
Number of attempts for the successful CBD cannulation | 3 hours
Overall cannulation success rate | 3 hours
complication rates | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No